CLINICAL TRIAL: NCT06423222
Title: Prevalence of Anal Incontinence and Its Impact on Quality of Life and Physical Activity Among Hungarian Women Who Have Given Birth, and the Hungarian Language Validation of the International Consultation on Incontinence Modular Questionnaire-Bowels (ICIQ-B)
Brief Title: Anal Incontinence and Its Impact on Quality of Life and Physical Activity Among Hungarian Women and the Hungarian Language Validation of the International Consultation on Incontinence Modular Questionnaire-Bowels (ICIQ-B)
Status: Recruiting | Type: Observational
Sponsor: University of Pecs (Other)
Responsible Party: Sponsor
Other Study IDs: BM/5814-3/2024
Record Dates: First submitted 2024-05-05; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Anal Incontinence
Keywords: Anal Incontinence; Quality of Life; Physical Activity; Questionnaire
MeSH Terms: conditions — Encopresis; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to assess the prevalence of anal incontinence among Hungarian women who have given birth at least once before, and to examine the impact of anal incontinence on the quality of life and physical activity of these women. A further aim of our study is to adapt the Hungarian version of the International Consultation on Incontinence Modular Questionnaire - Bowels (ICIQ-B) and to assess its validity and reliability.

ELIGIBILITY:
Inclusion Criteria:

* Have given birth at least once before
* Native Hungarian language

Exclusion Criteria:

* Menopause
* Irritable Bowel Syndrome (IBS)
* Chron's disease
* Ulcerative colitis
* Developmental abnormalities at the level of the pelvic organs
* Uninvestigated pelvic pain
* Malignant pelvic tumor
* Radiotherapy involving the pelvis
* Neurological diseases with muscle weakness
* Parkinson's disease
* Intellectual disability

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: We plan to include subjects who are female, over the age of 18, under the age of 50 and who have given birth at least once before.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Anal Incontinence Impact on Quality of Life | Through study completion, an average of 3 years
  Assessing with questionnaire: International Consultation on Incontinence Modular Questionnaire-Bowels (ICIQ-B). The ICIQ-B is a patient-completed questionnaire to assess the symptoms and impact on quality of life (QoL) of anal incontinence (including flatus incontinence). The ICIQ-B consists of 21 items, divided into three domains: Bowel pattern (1 - 21), bowel control (0 - 28), Quality of life (0 - 26). Seventeen items are scored items and the remaining four are unscored. Higher scores indicate more symptoms.
Anal Incontinence Impact on Physical Activity | Through study completion, an average of 3 years
  Assessing with questionnaire: Global Physical Activity Questionnaire (GPAQ). The Global Physical Activity Questionnaire was developed by WHO to monitor physical activity in countries. It collects information from 16 questions (P1-P16) on participation in physical activity in three domains (Workplace activity, Travel to and from places, Leisure activities) and sedentary behavior. Metabolic equivalent (MET) values are applied to the time variables according to the intensity of the activity (moderate or high). The application of MET values to activity levels allows the calculation of total physical activity.
Adaptation, validity and reliability of the Hungarian version of the International Consultation on Incontinence Modular Questionnaire-Bowels (ICIQ-B) | Through study completion, an average of 3 years
  Evaluating with statistical analysis the content/face validity, internal consistency, construct validity, test-retest reproducibility, discriminant validity and convergent validity.

SECONDARY OUTCOMES:
Additional pelvic floor symptoms | Through study completion, an average of 3 years
  Assessing with questionnaire: The Hungarian version of the Australian Pelvic Floor Questionnaire (APFQ-H). The APFQ-H consists of four domains: bladder function (15 items), bowel function (12 items), prolapse symptoms (5 items) and sexual function (10 items). Thirty-eight of the items assess pelvic floor symptoms and four questions assess the bother caused by symptoms in each domain. Most items in the questionnaire use a 4-point scoring system. The score obtained for each domain ranges from 0 to 10. The sum of the subscores in the four domains gives the APFQ-H global score. The higher the score, the more severe the pelvic floor symptoms.
Global Quality of Life | Through study completion, an average of 3 years
  Assessing with questionnaire: Hungarian WHOQOL-BREF. The WHOQOL-BREF is a self-administered questionnaire that contains 26 questions about an individual's health and well-being over the previous two weeks. Answers to the questions are given on a Likert scale of 1-5. The WHOQOL-BREF covers four domains (physical health, psychological, social relationships, environment). Scores in each of the 4 domains are converted into a scale ranging from 0 to 100. A score of 0 represents the worst possible health status, while a score of 100 represents the best possible health status for that domain.

CONTACTS AND LOCATIONS:
Overall Officials: Márta Hock, PhD, Study Director — University of Pécs Faculty of Health Sciences; Eszter Ambrus, Principal Investigator — Doctoral School of Health Sciences, Faculty of Health Sciences, University of Pécs, Pécs, Hungary
Locations (1):
- Doctoral School of Health Sciences, Faculty of Health Sciences, University of Pécs, Pécs, Baranya, Hungary

IPD SHARING:
Plan to Share IPD: No